CLINICAL TRIAL: NCT01300897
Title: Investigation of Cortico-Rectal Pathways in Healthy Subjects and Constipated Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Satish Rao, Professor, Augusta University
Other Study IDs: 5R01DK057100-2; 5R01DK057100 (NIH)
Record Dates: First submitted 2010-08-18; First posted 2011-02-23 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Healthy Volunteers; Constipation
Keywords: cortical evoked potentials, motor evoked potential responses
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy Volunteer: healthy volunteers will serve as controls. In each subject the cortical evoked potentials, transcranial motor evoked potentials and translumbosacral motor evoked potentials will be measured.
  Interventions: Procedure: Cortical Evoked Potentials; Procedure: Transcranial motor evoked potentials; Procedure: Translumbosacral motor evoked potentials
- Constipated patients: Patients with chronic constipation and rectal hypersensitivity or hyposensitivity and/or dyssynergic defecation.In each subject the cortical evoked potentials, transcranial motor evoked potentials and translumbosacral motor evoked potential will be measured
  Interventions: Procedure: Cortical Evoked Potentials; Procedure: Transcranial motor evoked potentials; Procedure: Translumbosacral motor evoked potentials

INTERVENTIONS:
Procedure: Cortical Evoked Potentials — A probe with 2 ring electrodes is placed in the anorectum. A small amount of electric current is passed separately through the anal and rectal electrodes.. The cortical evoked potentials from the anal and rectal sites are measured.
Procedure: Transcranial motor evoked potentials — A probe with 2 ring electrodes is placed in the anorectum. A magnetic coil is placed on the scalp at the anorectal site on each side, and discharged using magnetic energy. The motor evoked potentials at the anal and rectal sites are measured.
Procedure: Translumbosacral motor evoked potentials — A probe with 2 ring electrodes is placed in the anorectum. A magnetic coil is placed on the back at the lumbar plexus and sacral plexus levels and discharged using magnetic energy. The motor evoked potentials at the anal and rectal sites are measured.

SUMMARY:
Biofeedback therapy improves bowel symptoms and anorectal function in patients with dyssynergic defecation, however its mechanism of action is not known. The investigators hypothesize that biofeedback therapy enhances gut-brain-gut communication by altering cortical processing of information and improving cortically mediated neuromuscular function of the gut. However, in order to better understand these mechanisms in patients, the investigators need to examine and establish normative data and compare findings with healthy subjects. The investigators specific aims are to examine and evaluate the following 40 normal subjects; (1) To evaluate the afferent cortical evoked potentials in response to the electrical stimulation of the anorectum and (2) To evaluate the corticofugal tracts (efferent) by recording the anal and rectal electromyographic responses following noninvasive lumbosacral and transcranial magnetic stimulation.

DETAILED DESCRIPTION:
1. Cortical evoked potentials:A probe with 2 ring electrodes is placed in anus and rectum. A small amount of electrical current is passed. The cortical evoked responses to the anal and rectal electrical stimulation is measured from the scalp using a neurophysiology recorder.
2. Motor evoked potentials: A magnetic coil is placed on the scalp at the anorectal cortical site and discharged using magnetic energy. The anal and rectal motor evoked potentials are then measured using a probe with 2 ring electrodes.

ELIGIBILITY:
Inclusion criteria:

* Right-handed adults between ages 18 years and 99 years, who are free of bowel disorders or other medical illnesses.

Exclusion Criteria:

* Potential subjects with comorbid illnesses; severe cardiac disease, chronic renal failure or previous gastrointestinal surgery except cholecystectomy and appendectomy.
* Neurologic diseases e.g.; head injury, epilepsy, multiple sclerosis, strokes, spinal cord injuries.
* People who have metal in their skull or under the skull, or have metal in the back or hips.
* People who have a cardiac pacemaker, implanted defibrillator or medication pump.
* Impaired cognizance (mini mental score of < 15) and/or legally blind.
* Pregnant or likely to conceive during the course of the study. Women with potential for pregnancy must be willing to use contraceptive measures during the study.
* Previous pelvic surgery, rectocele repair, bladder repair, radical hysterectomy.
* Rectal prolapse or anal fissure or anal surgery.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 40 Healthy volunteers. 110 patients with chronic constipation and dyssynergic defecation and rectal hyposensitivity and rectal hypersensitivity
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2005-08 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Describe latencies and amplitudes between the brain and gut in healthy volunteers | 1 visit of 3 hours
  Measurements & Analysis: The latency, inter-peak latency and amplitude of each component of the cortical evoked potentials will be averaged to obtain group mean data.
  Statistical Analysis: The paired t-test or Wilcoxon signed-rank test will be used to compare the latencies.
  Lumbosacral and Transcranial Magnetic Stimulation (TMS) Data and Statistical Analysis: Mean latency and mean amplitude for each individual will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Satish SC Rao, MD, PhD, Principal Investigator — Augusta University
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States